CLINICAL TRIAL: NCT02031120
Title: Improved Management Based on Pathophysiology of Drug Hypersensitivity in Childhood
Brief Title: Management of Drug Hypersensitivity in Children
Acronym: DHC
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting participants.
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Christoph Caubet, Chef de clinique, University Hospital, Geneva
Other Study IDs: UGeneva 13-006
Record Dates: First submitted 2014-01-05; First posted 2014-01-09 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Drug Hypersensitivity
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is (1) to assess the incidence of suspected drug allergies in a pediatric hospital and the proportion in which these reactions are confirmed to be allergic; (2) to evaluate the diagnostic values of the different allergy tests available; (3) to investigate the pathophysiology of drug allergies, particularly by investigating the role of viruses, and by performing HLA typing and a gene expression profile both in the acute phase of the reaction and 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* Participation will be proposed to any children (0 to 16 years) receiving one or several drug(s) and developing one of the following clinical manifestations: urticaria, maculopapular rash, bullous eruption, flush, anaphylaxis, serum sickness-like disease, SJS, TEN, DRESS or fever linked to drug intake.

Exclusion Criteria:

* Patients will be excluded if the symptoms occur more than 72 hours after any treatment was stopped or if the symptoms are clearly linked to another cause (measles, rubeola, roseola, varicella, fifth disease, Gianotti-Crosti syndrome, scarlet fever, Gibert's pityriasis or food allergy).

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with suspected drug allergies in a pediatric hospital (including ambulatory departments)
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of suspected drug allergies in a pediatric hospital and the proportion in which these reactions are confirmed to be allergic | 3 years

SECONDARY OUTCOMES:
Evaluation of the diagnostic values of the different allergy tests available | 3 years
  Sensitivity, specificity, negative and positive predictive value
Determination of the role of viruses, HLA typing and gene expression profile both in the acute phase of the reaction and 2 months later | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christoph Caubet, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland